CLINICAL TRIAL: NCT00080795
Title: Phase II Trial of Neoadjuvant, Multi-Agent Chemotherapy For Locally Advanced Urothelial Cancer
Brief Title: Neoadjuvant Ifosfamide, Doxorubicin, Gemcitabine, and Cisplatin in Treating Patients Who Are Undergoing Radical Cystectomy for Locally Advanced Carcinoma (Cancer) of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000355361; MDA-ID-01317; ID01-317 (Other: UT MD Anderson Cancer Center)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: stage III bladder cancer; regional transitional cell cancer of the renal pelvis and ureter; anterior urethral cancer; posterior urethral cancer; urethral cancer associated with invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Filgrastim; Cisplatin; Doxorubicin; Gemcitabine; Ifosfamide; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: gemcitabine hydrochloride
Drug: ifosfamide
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ifosfamide, doxorubicin, gemcitabine, and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug, and giving them before surgery, may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well neoadjuvant combination chemotherapy works in treating patients undergoing radical cystectomy for locally advanced carcinoma of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate and 4-year disease-free survival of patients with locally advanced carcinoma of the urothelium undergoing radical cystectomy treated with neoadjuvant chemotherapy comprising ifosfamide, doxorubicin, and gemcitabine followed by cisplatin, gemcitabine, and ifosfamide.

Secondary

* Compare perioperative morbidity and mortality of patients treated with this regimen vs historical standards.

OUTLINE: Patients receive neoadjuvant chemotherapy comprising ifosfamide IV over 3 hours on days 1-4, doxorubicin IV on day 3, gemcitabine IV over 30 minutes on days 2 and 4, and filgrastim (G-CSF) subcutaneously on days 7-12 or until blood counts recover. Treatment repeats every 3 weeks for a total of 3 courses. Patients then receive cisplatin IV, gemcitabine IV over 90 minutes, and ifosfamide IV over 30 minutes on day 1. Treatment repeats every 2 weeks for a total of 4-6 courses. Four to six weeks after the completion of all neoadjuvant chemotherapy, patients undergo cystectomy.

Patients are followed at 9, 12, 15, 18, 24, and 30 months and then annually thereafter.

PROJECTED ACCRUAL: A total of 31-49 patients will be accrued for this study within 16-25 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the urothelium, meeting 1 of the following criteria for locally advanced disease:

  * Clinical stage T3b disease, defined by presence of a mass on examination under anesthesia
  * Clinical stage T4a disease, defined by direct invasion of prostatic stroma, vagina, or rectum
  * Lymphovascular invasion on transurethral resection specimen
* Upper tract disease or micropapillary histology allowed
* No evidence of disease outside the pelvis

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* 0-2

Life expectancy

* Not specified

Hematopoietic

* Bone marrow function adequate

Hepatic

* Liver function adequate

Renal

* Creatinine clearance ≥ 45 mL/min

Cardiovascular

* Ejection fraction ≥ 50%

Other

* Not pregnant
* No other malignancy likely to be life-threatening within the next 4 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2001-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 weeks following treatment
Disease-free survival at 4 years | 4 years

SECONDARY OUTCOMES:
Comparison of perioperative treatment morbidity and mortality with historical standards | Minimally reviewed following 6 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Randall E. Millikan, MD, PhD, Study Chair — M.D. Anderson Cancer Center; Colin P. Dinney, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center at University of Texas, Houston, Texas, United States